CLINICAL TRIAL: NCT01139619
Title: A Retrospective, Medical Record Study to Investigate the Current Situation of Biopsy Testing in the Swedish Inoperable Non Small Cell Lung Cancer Patient Population
Brief Title: A Retrospective Study to Investigate the Current Situation of Biopsy Testing in Swedish Inoperable Non Small Cell Lung Cancer (NSCLC) Patients
Acronym: MAPSY
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OSE-DUM-2010/1
Record Dates: First submitted 2010-06-02; First posted 2010-06-08 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Biopsy Mapping; Non small cell lung cancer; NSCLC; Lung cancer diagnosis; Retrospective; Inoperable Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Inoperable non small cell lung cancer patients. Diagnosed between 2010-05-31 and 2009-06-01.

SUMMARY:
Lung cancer is one of the most deadly types of cancer and the leading cause of death in cancer in Sweden. Five year survival is 10% in men and 15% in women. Approximately 3300 individuals in Sweden are diagnosed each year and the incidence of adenocarcinoma is increasing. Lung cancer patients are to a great extent currently being diagnosed by exfoliative cytology. However, new drugs leading to more personalized treatments will demand more specific classification of tumour types. Today EGFR mutation status is becoming an important factor when deciding treatment strategy for patients with Non-Small Cell Lung cancer.

Sufficient tumour material must be available if EGFR mutation status is to be tested. Core needle biopsy is one way to obtain the quantity of material needed when testing mutation status. The portion of patients having core needle biopsies is believed to vary greatly between hospitals in Sweden, a difference from 20% to 70 % have been assumed, but is not yet confirmed in studies. This study will investigate the current situation and procedures when patients are diagnosed with lung cancer. The results can be used to describe any possible adverse events connected to the procedure and possibly contribute to development of a better decision tool to be used when deciding if a core needle biopsy is to be performed or not.

More and more therapeutical targets having similar problems are likely to be developed in the future. An investigation of current quality and procedures when diagnosing lung cancer by biopsies will facilitate future diagnosing of lung cancer and ensure that personalized treatments can be offered to patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis code C34 (ICD-10).
* Inoperable lung cancer.
* Diagnosis of lung cancer made between 2010-05-31 and 2009-06-01.

Exclusion Criteria:

* Diagnosis code C34.9b.
* Diagnosis code C34.9h.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 200 inoperable non small cell lung cancer patients recruited from centers in Swedish University- and County hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Describe complications connected to biopsy and bronchoscopy in the investigated lung cancer population. | Data will be collected retrospectively from medical records. Data of complications will be collected from when the complication occurred and then any overnight stay caused by complication, approximately a few days.
Describe time to diagnosis for patients diagnosed by transthoracic biopsy compared to patients diagnosed by bronchoscopy. | Data will be collected retrospectively from medical records. The time span assessed will be from first contact at hospital to the date of diagnosis. Approximately a time frame of a few weeks up to several months.
Describe difference in clinical outcome for patients diagnosed by histopathology compared to patients diagnosed by cytology alone, one year after diagnosis. | Data will be collected retrospectively from medical records. The time of data collection will be at least one year after diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Pål Falck, PhD, Study Director — AstraZeneca; Hirsh Koyi, MD PhD, Principal Investigator — Gävle Hospital
Locations (3):
- Sweden (3):
  - Research Site, Gävle
  - Research Site, Linköping
  - Research Site, Luleå